CLINICAL TRIAL: NCT00813553
Title: Effect of Two 8-week β-alanine Supplementation Protocols on Muscle Carnosine
Brief Title: Effect of β-alanine Supplementation on Muscle Carnosine
Acronym: LitmusMagnet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: University of Bern (Other); Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 08.13.PER
Record Dates: First submitted 2008-12-22; First posted 2008-12-23 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Healthy
Keywords: physical fitness; exercise; amino acid
MeSH Terms: conditions — Motor Activity | interventions — beta-Alanine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- beta-alanine 0 (Placebo Comparator)
  Interventions: Dietary Supplement: placebo
- beta-alanine 1 (Experimental)
  Interventions: Dietary Supplement: beta-alanine
- beta-alanine 2 (Experimental)
  Interventions: Dietary Supplement: beta-alanine

INTERVENTIONS:
Dietary Supplement: placebo — daily
  Arms: beta-alanine 0
Dietary Supplement: beta-alanine — daily
  Arms: beta-alanine 1
Dietary Supplement: beta-alanine — daily
  Arms: beta-alanine 2

SUMMARY:
Carnosine is a natural acid buffering substance of muscle. The primary objective of this study is to test whether a nutritional supplement of beta-alanine enhances carnosine content in muscle.

DETAILED DESCRIPTION:
Volunteers will be randomized to receiving 3 nutritional supplements. Two supplements contain beta-alanine at different doses, the third supplement is a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Stable health as evaluated by medical evaluation
* Body mass index higher than 18 kg/m2
* Body mass index lower than 25 kg/m2, unless body fat is less than 20%

Exclusion Criteria:

* intolerance to β-alanine,
* allergy to soy, fish and crustacean
* participation in another intervention study
* consumer of dietary supplement susceptible to contain beta-alanine
* determined to have very high baseline muscle carnosine concentration

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
muscle carnosine concentration | 0 to 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University and Inselspital, Bern, Canton of Bern, Switzerland